CLINICAL TRIAL: NCT05039463
Title: Efficacy at One Year of Combined Injections of Plasma Rich in Platelets and Hyaluronic Acid in Knee Osteoarthritis
Acronym: ISPAG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2021_843_0178
Record Dates: First submitted 2021-08-31; First posted 2021-09-09 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Knee Osteoarthritis; Hyaluronic Acid; Platelet Rich Plasma
Keywords: platelet rich plasma; hyaluronic acid; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PRP + HA: two injections of PRP (plasma rich in platelets ), in combination with HA (hyaluronic acid)
- HA alone: HA (hyaluronic acid)

SUMMARY:
The French Society of Rheumatology cannot rule on the value of intra-articular injections of PRP due to the lack of hindsight and insufficient data. In fact, the injection protocols are very heterogeneous in terms of preparation method, the presence or not of leukocytes, the number of centrifugations, the volume injected, the ultrasound guidance, which makes it difficult to analyze the literature. The investigator objective is therefore to evaluate the effectiveness of combined injections of PRP and hyaluronic acid.

ELIGIBILITY:
Inclusion Criteria:

* age : > 18 years old
* Patients benefiting, in the context of knee osteoarthritis, from viscosupplementation alone or from two injections of PRP, in combination with HA, at the Amiens University Hospital.

Exclusion Criteria:

* Patient refusal to use the data
* Language barrier
* Age less than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients benefiting, in the context of knee osteoarthritis, from viscosupplementation alone or from two injections of PRP, in combination with HA, at the Amiens University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
change of the visual analogue scale (VAS) from the "PRP + HA" group on the "HA alone" group | up to one year

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No